CLINICAL TRIAL: NCT03867682
Title: A Phase I/II Study of Venetoclax and Lintuzumab-Ac225 in Patients With Refractory or Relapsed AML
Brief Title: Venetoclax and Lintuzumab-Ac225 in AML Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Actinium Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LIN-AC225-AML02
Record Dates: First submitted 2019-03-06; First posted 2019-03-08 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Acute Myeloid Leukemia; Relapsed Adult AML
Keywords: Lintuzumab-Ac225; Venetoclax; Lintuzumab; Refractory AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Spironolactone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase I and Phase II (Experimental): Lintuzumab-Ac225 administered on Day 5 of each cycle for four cycles (unless in the 0.5 μCi/kg or 0.25 μCi/kg cohorts, where there is a potential for an additional four cycles, pending PI and Medical Monitor review).
  Venetoclax taken on Days 1-21 of each cycle for up to 12 cycles.
  Each cycle is 28 days, with a potential to expand to 42 days to allow for full hematologic recovery.
  Interventions: Biological: Lintuzumab-Ac225; Drug: Venetoclax; Drug: Spironolactone

INTERVENTIONS:
Biological: Lintuzumab-Ac225 — In the Phase I, patients will be enrolled into the following dose escalation cohorts: 0.50 μCi/kg, 1.0 μCi/kg, and 1.5 μCi/kg. If the 0.50 μCi/kg dose is determined to exceed the MTD, a 0.25 μCi/kg dose will be explored.
  Other Names: Actimab
Drug: Venetoclax — 400 mg daily will be taken orally on Days 1-21 of a 28-day cycle. There will be a ramp up of venetoclax dosing in the first cycle, with 100 mg administered on Day 1, 200 mg on Day 2, and 400 mg on Day 3 and Day 4 and later. Patients on antifungal azoles should receive one-half these doses, up to a maximum of 200 mg of venetoclax.
  Other Names: Venclexta
Drug: Spironolactone — 25 mg by mouth daily, administered on Cycle 1 Day 15 and continued for 12 months after the subject's last treatment with lintuzumab-Ac225.
  Other Names: Aldactone

SUMMARY:
The study is a multicenter, open label Phase I/II trial.

1. To determine the maximum tolerated dose (MTD) of lintuzumab-Ac225 added to venetoclax for patients with CD33 positive relapsed/refractory AML. (Phase 1 portion)
2. To assess the percentage of patients with CR, CRh, or Overall Response (CR + CRh), up to 6 months after the start of treatment without receiving other AML therapies. (Phase 2 portion)

DETAILED DESCRIPTION:
The study is a multicenter, open label Phase I and Phase II trial combining lintuzumab-Ac225 with venetoclax in patients who have relapsed or refractory AML.

The Phase I portion is a dose-finding study which will enroll at least three patients at each dose level. Patients in a dose level will be observed for a minimum of 4 weeks before dose escalation occurs. There is no dose escalation for any individual patient.

The Phase II portion of the study will enroll patients at the MTD dose level of lintuzumab-Ac225 as determined in the Phase I portion of the study. The goal of the Phase II portion will be to further characterize the safety and efficacy of the MTD dose of lintuzumab-Ac225.

ELIGIBILITY:
Inclusion Criteria:

1. Refractory or relapsed AML which will include:

   1. Refractory disease will be defined as at least 1 prior treatment with no remission.
   2. Relapsed disease will be defined as 5% or more blasts in bone marrow seen after remission.
   3. Patients with AML arising from myelodysplastic syndromes (including CMML) or myeloproliferative neoplasms (secondary AML, ts-AML) are also eligible.
2. Circulating blast count ≤ 200/μL within 10 days prior to first cycle of treatment. Hydroxyurea should be used to keep the peripheral blast count ≤ 200/μL until the first day of protocol treatment, to the extent that this is possible
3. ECOG ≤ 2
4. Estimated creatinine clearance ≥ 50 mL/min
5. AST and ALT ≤ 3.0 x ULN
6. Bilirubin ≤ 3.0 x ULN

Exclusion Criteria:

1. Active CNS Leukemia.
2. Known HIV infection or known hepatitis B or hepatitis C infection (with a detectable viral load).
3. Participant has received strong and/or moderate CYP3A inducers within 7 days prior to the initiation of study treatment.
4. Secondary refractory AML (e.g., treated for current relapse without achieving remission);

   a. With the exception that single agent FLT3 inhibitors, IDH1/IDH2 inhibitors are allowed for current relapse without achieving remission.
5. Have received prior radiation to maximally tolerated levels to any critical normal organ.
6. Clinically significant cardiac disease.
7. Active, uncontrolled serious infection.
8. Have other non-myeloid malignancy within 2 years of entry (with exceptions).
9. Psychiatric disorder that would preclude study participation
10. Previous solid organ transplant (prior treatment with SCT is allowed but not if patient has GVHD or is still receiving immunosuppression/GVHD therapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2020-01-15 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Phase I: Maximum Tolerated Dose (MTD) of Lintuzumab-Ac225 | Cycle 1, up to 48 days
  To determine the maximum tolerated dose (MTD) of lintuzumab-Ac225 added to venetoclax for patients with CD33 positive relapse/refractory AML.
Phase II: Overall Response (CR + CRh + CRi) | Up to 6 months
  To assess the percentage of patients with CR, CRh, CRi or Overall Response (CR + CRh + CRi), up to 6 months after the start of treatment without receiving other AML therapies.

SECONDARY OUTCOMES:
Phase I: Overall Response | Up to 6 months
  Number of patients who's overall response is CR, CRh, or CRi
Phase I and II: OS | End of 6 months, 12 months, 2 years
  Number of patients who died
Phase I and II: DFS | End of 6 months, 12 months, 2 years
  Disease-free survival
Phase I and II: Evaluate incidence of AEs and SAEs | Through study completion, up to 2 years
  Rate of AEs and SAEs, including infusion-related reactions
Phase I and II: Evaluate BH3 priming assay results | Completion of Cycle 1, estimated 1 month
  Summary of assay results
Phase I and II: MRD status | From date of first dose until the date of first documented response, first assessment at 6 months
  Number of patients who are MRD negative
Phase I and II: Lab abnormalities (other than hematologic indices) | Through study completion, up to 2 years
  Summary of rate of Grade 3/4 lab abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Avinash Desai, MD, Study Chair — Actinium Pharmaceuticals, Inc.
Locations (5):
- United States (5):
  - University of California, Los Angeles, California
  - University of Louisville, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Weill Cornell Medicine, New York, New York
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- [Derived] Garg R, Allen KJH, Dawicki W, Geoghegan EM, Ludwig DL, Dadachova E. 225Ac-labeled CD33-targeting antibody reverses resistance to Bcl-2 inhibitor venetoclax in acute myeloid leukemia models. Cancer Med. 2021 Feb;10(3):1128-1140. doi: 10.1002/cam4.3665. Epub 2020 Dec 21. PMID 33347715